CLINICAL TRIAL: NCT05539560
Title: The Effect of Olfactory Training in Patients With COVID-19 Induced Olfactory Dysfunction - A Randomized Placebo-controlled Clinical Trial
Brief Title: The Effect of Olfactory Training in Patients With COVID-19 Induced Olfactory Dysfunction
Acronym: SMELLT2022
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ditte Gertz Mogensen (Other)
Responsible Party: Sponsor-Investigator, Ditte Gertz Mogensen, PhD-student, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-ENT-1-olfactory
Record Dates: First submitted 2022-09-02; First posted 2022-09-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: Olfactory training; Quality of life; Olfactory dysfunction; Covid-19; Parosmia
MeSH Terms: conditions — COVID-19; Olfaction Disorders | interventions — Olfactory Training; Oils, Volatile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Olfactory training twice a day with essential oils
  Interventions: Other: Olfactory training with essential oils
- Control group (Placebo Comparator): Olfactory training twice a day with fragrance-free oils
  Interventions: Other: Olfactory training with fragrance-free oils

INTERVENTIONS:
Other: Olfactory training with essential oils — Olfactory training twice daily with essential oils from Urtegaarden Aps with scents of orange, lavender, clove and peppermint. The olfactory training is performed every morning and evening, by smelling each of the oils for 30 seconds.
  Other Names: Urtegaarden ApS Essential Oils
  Arms: Intervention group
Other: Olfactory training with fragrance-free oils — Olfactory training twice daily with fragrance-free oils from Urtegaarden Aps in the same four containers as the intervention group. The olfactory training is performed every morning and evening, by smelling each of the oils for 30 seconds.
  Other Names: Urtegaarden ApS Essential Oils (Fragrance-free custom made)
  Arms: Control group

SUMMARY:
Aim: The aim is to investigate the effect of olfactory training with essential oils versus olfactory training with placebo-oils in patients with COVID-19 induced olfactory dysfunction

Study design: The study is a placebo-controlled randomized clinical trial with an intervention group and a control group. The intervention group receive four essential oils with scents of orange, lavender, clove, and peppermint. Patients in the control group receive a fragrance kit, consisting of the same containers, but with fragrance-free oils added. Both groups are instructed to smell each of the four oils for 30 seconds in the morning and evening, over a three-month intervention period. Patients are given a diary in which to record their olfactory training. The nurse or medical student instructing the patients in the training and performing the smell and taste tests is blinded.

Study population: Patients referred to the Unit for Sense of Taste and Smell in the Department of Otorhinolaryngology Head & Neck and Audiology at Rigshospitalet.

Inclusion criteria:

* Impaired sense of taste and smell following COVID-19 > 3 months
* Hyposmia (16.25-30.5) or anosmia (<16) assessed by Sniffin' Sticks Olfactory Test for Threshold, Discrimination and Identification (TDI) performed in the Unit for Sense of Taste and Smell with or without parosmia based on medical history
* > 18 years of age

Exclusion criteria:

* Cause of hyposmia, anosmia or parosmia other than COVID-19
* Does not read or speak Danish
* Lack of compliance to perform daily olfactory training

Procedures:

- TDI-test: To assess patients' sense of smell, the TDI-test with Sniffin' Sticks is used, which is a validated tool with normative data.

Questionnaires:

- 'Taste and Smell Tool for Evaluation' is used to investigate quality of life related to impaired sense of taste and smell.

ELIGIBILITY:
Inclusion Criteria:

* Olfactory dysfunction caused by COVID-19
* Hyposmia (16.25-30.5) or anosmia (<16) with or without parosmia assessed by TDI test with Sniffin Sticks performed in the Unit for Sense of Taste and Smell
* > 18 years of age

Exclusion Criteria:

* Cause of hyposmia, anosmia or parosmia other than COVID-19
* Does not read or speak Danish
* Lack of compliance to perform daily olfactory training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Extended Sniffin' Sticks Test score | 3 months follow-up
  Change in TDI score measured by Burghart Extended Sniffin' Sticks Test (TDI test). The TDI test, consists of a threshold test, a discrimination test, and an identification test. The results of the three subtests makes a total TDI score, where the minimum score is 1 and the maximum score is 48. A score >30 indicates normal olfactory function, a score between 15-30 indicates hyposmia and a score <15 indicates anosmia in the form of severely impaired or complete loss of olfaction.

SECONDARY OUTCOMES:
Change in Quality of Life | 3 months follow-up
  Change in Quality of Life measured by the questionnaire Taste and Smell Tool for Evaluation. The minimum score is 21 and the maximum score is 105. A higher score means worse outcome (quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke G Backer, Professor, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Mogensen DG, Aanaes K, Andersen IB, Jarden M, Backer V. Effect of Olfactory Training in COVID-19 Related Olfactory Dysfunction-A Placebo-Controlled Trial. Laryngoscope. 2025 Dec;135(12):4849-4857. doi: 10.1002/lary.32275. Epub 2025 May 15. PMID 40371997

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT05539560/Prot_SAP_ICF_000.pdf